CLINICAL TRIAL: NCT02088333
Title: A Primary Care Multilevel mHealth Colorectal Cancer Screening (mCRC) Intervention
Brief Title: Effectiveness of an mHealth Colorectal Cancer Screening Intervention
Acronym: mCRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00023575; 1R01CA178941 (NIH); CCCWFU 59A13 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer screening; computer-assisted instruction; mHealth; text message
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mCRC intervention (Experimental): intervention arm
  Interventions: Behavioral: mCRC intervention
- Healthy lifestyles education (Placebo Comparator): tablet-based patient education about healthy lifestyles
  Interventions: Behavioral: Healthy Lifestyles video

INTERVENTIONS:
Behavioral: mCRC intervention — a multilevel intervention consisting of tablet-based patient education about CRC screening, post-visit patient electronic messaging, and clinic protocols to facilitate ordering of screening tests
  Arms: mCRC intervention
Behavioral: Healthy Lifestyles video — a brief video about healthy lifestyle habits displayed on a tablet device
  Arms: Healthy lifestyles education

SUMMARY:
The purpose of this study is to determine whether a multilevel mHealth intervention (mCRC) can increase the percentage of patients who receive colorectal cancer screening. The mCRC intervention will include a tablet-based patient education program, clinic protocols to facilitate the ordering of CRC screening tests, and electronic messaging with patients to promote screening. The investigators hypothesize that participants randomized to mCRC will be more likely to complete screening compared with those randomized to the control arm of the study. Additionally, the investigators hypothesize mCRC will increase several intermediate outcomes (such as knowledge, attitudes, beliefs, and test ordering) which will predict completion of screening. Lastly, the investigators hypothesize the mCRC intervention will add little to the overall cost of screening.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients aged 50 - 74 years
* Scheduled to see a primary care provider for a routine (i.e., non-urgent care) visit
* Due for colorectal cancer screening

Exclusion Criteria:

* A personal history of CRC
* Specific CRC risk factors, including: First degree relative with CRC; Personal history of adenomatous polyps; Recent blood in stools
* Obvious physical or mental disability that would prevent participant from interacting with a tablet device.
* Receipt of treatment for cancer (excluding non-melanoma skin cancers) within the last 6 months.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Completion of CRC Screening | 24 weeks
  Patient completion of a colorectal cancer screening test, such as the fecal occult blood test, a flexible sigmoidoscopy, or a colonoscopy.

SECONDARY OUTCOMES:
CRC Screening Attitudes and Beliefs | Day of enrollment
  A survey scale measuring the participant's attitudes and beliefs about CRC screening
Intention to receive CRC screening | Day of enrollment
  Participant's stated intention to receive CRC screening
Self-efficacy | Day of enrollment
  Participant's belief that they are capable of completing CRC screening
Ability to make a screening decision | Day of enrollment
CRC screening discussions | Up to 5 days
  Participants' self-report of whether they discussed CRC screening with a medical provider
Satisfaction with screening decision | Up to 5 days
  Survey questions based on the Satisfaction with Decision Scale
CRC screening test order | 24 weeks
  Whether or not a CRC screening test was ordered for the participant
Cost of the mCRC intervention | 24 weeks
  Additional cost of the mCRC intervention as captured by additional time and technology costs
Usability of the mCRC system | Day of enrollment
  Participant's rating of the usability of the mCRC system

CONTACTS AND LOCATIONS:
Overall Officials: David P Miller, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Hillsdale Family Medicine, Advance, North Carolina
  - Foothills Family Medicine, Mount Airy, North Carolina
  - Wilkes Internal Medicine, Wilkesboro, North Carolina
  - Downtown Health Plaza, Winston-Salem, North Carolina
  - Peace Haven Family Medicine, Winston-Salem, North Carolina
  - Reynolda Family Medicine, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Miller DP Jr, Denizard-Thompson N, Weaver KE, Case LD, Troyer JL, Spangler JG, Lawler D, Pignone MP. Effect of a Digital Health Intervention on Receipt of Colorectal Cancer Screening in Vulnerable Patients: A Randomized Controlled Trial. Ann Intern Med. 2018 Apr 17;168(8):550-557. doi: 10.7326/M17-2315. Epub 2018 Mar 13. PMID 29532054